CLINICAL TRIAL: NCT07073924
Title: Prescribe to Prevent HIV (P2PH): Enhancing Clinic-based Prescribing of Harm Reduction: A Clinical Trial to Prevent HIV and Severe Injection-related Infections Among PWID
Brief Title: Prescribe to Prevent HIV: A Hybrid Trial Helping Addiction Clinics Prevent HIV & Infections Through Safer Drug Use Support
Acronym: P2PH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Raagini Jawa, Assistant Professor of Medicine, University of Pittsburgh
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY25050118; K23DA063654 (NIH)
Record Dates: First submitted 2025-07-16; First posted 2025-07-20 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-07

CONDITIONS: People Who Use Opioids/People With Opioid Use Disorder (OUD)
Keywords: people who use drugs; HIV; PrEP; Opioid-Related Disorders; implementation; Substance-Related Disorders
MeSH Terms: conditions — Opioid-Related Disorders; Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: Cluster randomized, waitlist-controlled hybrid type 3 implementation-effectiveness pilot trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Arm (Other): Immediately gets the intervention of the implementation strategy bundle.
  Interventions: Behavioral: Implementation strategy bundle
- Waitlist Control Arm (Other): Waits for 6 months with no intervention, then gets the intervention of the implementation strategy bundle.
  Interventions: Behavioral: Implementation strategy bundle

INTERVENTIONS:
Behavioral: Implementation strategy bundle — The anticipated strategy bundle will include integrated patient-, provider-, and system-level interventions to support sustainable implementation. At the patient level, this may involve education, peer support, and navigation services; at the provider level, training, decision-support tools, and workflow enhancements; and at the system level, policy changes, electronic health record integration, and organizational alignment to promote and maintain prescribing of PrEP and injection equipment.

SUMMARY:
In the U.S., an estimated 3.6 million people who inject drugs (PWID) face a growing yet preventable health crisis, with rising cases of serious injection-related infections (SIRI), including HIV, due to limited access to two high-priority interventions: sterile injection equipment and daily oral HIV pre-exposure prophylaxis (PrEP). Outpatient clinics represent an opportune venue to implement these interventions. Yet most clinical providers in these settings do not currently provide them, contributing to a wide gap between evidence and routine practice. The Prescribe to Prevent HIV (P2PH) trial is a participatory study designed to co-develop and pilot test a set of implementation strategies to support outpatients clinics in offering sterile injection equipment and PrEP with the goal of reducing the risk of HIV and SIRI among PWID.

DETAILED DESCRIPTION:
In the U.S., 3.6 million people who inject drugs (PWID) face a syndemic of overdose and severe injection related infections (SIRI). Current efforts addressing this crisis remain inadequate as evidence-informed interventions (EIIs) to prevent or reduce SIRI from injection opioid use are not widely implemented and typically limited to syringe service programs. SIRI, which includes bacterial infections (e.g., cellulitis, osteomyelitis, endocarditis), hepatitis C virus, and HIV, significantly increase morbidity, mortality, and costs. HIV, in particular, can be prevented through access to two EIIs: sterile injection equipment and pre-exposure prophylaxis (PrEP). However, PWID in many jurisdictions lack access to these interventions due to shortages of syringe servie programs and clinicians willing to prescribe them. As a result, PWID nationwide have seen rising HIV incidence, threatening the goal of ending the HIV epidemic by 2030. For example, in Pennsylvania, where 90% of PWID lack access to SSPs, acute HIV infections rose by 150% between 2016 and 2019, and SIRI-related hospitalizations increased by 250% since 2010. This wide evidence-to-implementation gap underscores the urgent need for participatory implementation research to integrate these two high-priority EIIs into routine medical practice.

Outpatient clinics represent a missed opportunity to implement these two EIIs. Outpatient clinics, including primary care and Federally Qualified Health Centers, are more accessible and face fewer restrictions than SSPs. While integrating these EIIs in outpatient clinics aligns with federal priorities, prescribing remains uncommon even in addiction treatment contexts. Modeling shows that when outpatient clinics prescribe injection equipment, SIRI-related hospitalizations are reduced by 30%, and when PrEP is prescribed, it increases uptake among PWID. However, gaps remain in how to effectively implement the prescribing of injection equipment and PrEP in these settings.

Prescribe to Prevent HIV, is a participatory study designed to co-create and pilot a tailored implementation strategy bundle for prescribing injection equipment and PrEP in four Pennsylvania Centers of Excellence in Opioid Use Disorders (COEs). The approach combines implementation science with human-centered design, engaging a collaborative of individuals with lived experience, clinicians, and organizations serving PWID throughout all study phases to ensure relevance and sustainability.

Development of the strategy bundle will begin by identifying implementation barriers and facilitators through 24 semi-structured interviews with COE patients, administrators, clinicians, and staff, guided by the Consolidated Framework for Implementation Research and informed by input from a community collaborative of individuals with lived experience. Then, using a human-centered design process, a tailored, practical, and adaptable strategy bundle will be co-created based on findings from the semi-structured interviews, insights from the community collaborative, and input gathered through four focus groups-one each with COE patients, clinicians, staff, and administrators-for implementation across the four COE sites.

A cluster randomized, waitlist-controlled hybrid type 3 implementation-effectiveness pilot trial will then be conducted at the 4 COEs. The trial will assess implementation of the strategy bundle for prescribing injection equipment and PrEP in outpatient clinics. Primary implementation outcomes will include site-level adoption and maintenance, measured by the proportion of clinicians prescribing injection equipment and/or PrEP at the end of the 6-month implementation period (adoption), and at 12 months (maintenance). Secondary outcomes will include patient-level SIRI-related hospitalizations and negative HIV test results.

ELIGIBILITY:
Patients:

Pre-implementation interviews (N=12), pre-implementation focus groups (N=8), and post-implementation interviews (N=10)

Inclusion Criteria:

-Adult patients with history of active injection drug use in the past 1 year from the 4 COEs

Exclusion Criteria:

* Ages <18
* If history of injection drug use >1 year
* Non-English speaking
* Pending or legal action that could prohibit or interfere with participation (Ie. incarceration)
* Residence or discharge to a treatment facility that bans the possession of drug checking supplies
* Acute, severe psychiatric condition in need of immediate treatment.

Clinical Partners:

Pre-implementation interviews (N=12), pre-implementation focus groups (N = 24), post-implementation surveys (N = 80), and post-implementation interviews (N=10)

Inclusion Criteria:

-Prescribing clinicians (e.g., physicians, advanced practice providers such as nurse practitioners and physician assistants), administrators, medical assistants, and nurses from the 4 COEs

Exclusion Criteria:

* Individuals not affiliated with the 4 COEs.
* Staff outside the specified roles (i.e., not prescribing clinicians, administrators, medical assistants, or nurses).
* Students, trainees, or individuals not credentialed in the eligible roles.
* Those on extended leave or not actively working during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 536 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Implementation Outcomes: Site Level Adoption | 6 months post implementation
  This is defined as the proportion of clinicians who prescribed injection equipment and/or PrEP per site, assessed at 6 months post-implementation, respectively using electronic health record data.
Implementation Outcomes: Site-level maintenance | 12 months post implementation
  This is defined as the proportion of clinicians who prescribed injection equipment and/or PrEP per site, assessed at 12 months post-implementation respectively using electronic health record data.
Implementation Outcomes: Acceptability of the strategy bundle | 6 months post implementation
  Acceptability of the implementation strategy bundle will be assessed via post-implementation surveys of participating clinical partners (N=60-80) using a reliable 4-item survey from Weiner et al., where scores ≥16 indicate "acceptable" if 80% of participants agree.

SECONDARY OUTCOMES:
Clinical Outcome: Rate of SIRI-related hospitalizations | 6 months pre-implementation and 6 months post-implementation
  We will assess the rate of SIRI-related hospitalizations by extracting electronic health record data from participating sites using an established search algorithm that identifies relevant cases through ICD-10 codes associated with injection drug use infections.
Clinical Outcome: Rate of negative HIV tests | 6 months pre-implementation and 6 months post-implementation
  We will assess the rate of negative HIV screening tests by extracting electronic health record data from participating sites using which will be collected as part of routine clinical care.

CONTACTS AND LOCATIONS:
Overall Officials: Raagini Jawa, MD, MPH, Principal Investigator — University of Pittsburgh
Locations (4):
- United States (4):
  - Latterman Family Health Center, Pittsburgh, Pennsylvania
  - Center for Psychiatric And Chemical Dependency Services, Pittsburgh, Pennsylvania
  - Internal Medicine Recovery Engagement Program, Pittsburgh, Pennsylvania
  - UPMC Magee-Womens Hospital, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Study protocol and statistical analysis plan for the primary outcomes will be published in a manuscript. Analytic code and participant-level data can be requested from Principal Investigators. Analysis files will be constructed from the stored electronic data and will be stripped of identifying information. Specifically, participants will be identified with a numeric identifier that is not related to any element of their personal identifying information.
Supporting Information: Study Protocol
Access Criteria: Data will only be shared with external investigators when a data use agreement (DUA) is executed between University of Pittsburgh and the requester's institution. The DUA will specify the requested data elements (each of which must be justified), the specific research question, the timeline for the project, and schedule for data.